CLINICAL TRIAL: NCT00203112
Title: A Multi-Centered, Randomized, Double-Blind, Placebo-Controlled, Parallel Study Assessing the Add-on Effect of Minocycline in Relapsing-Remitting Multiple Sclerosis (RR-MS) Subjects Treated With Glatiramer Acetate (GA).
Brief Title: Safety and Efficacy Study of Copaxone Administered in Combination With Minocycline
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Jean-Louis Strill, MD, Teva Canada Innovation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GA 9014
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2011-04-12 (Estimated); Status verified 2011-04

CONDITIONS: Relapse Remitting Multiple Sclerosis
MeSH Terms: interventions — Glatiramer Acetate; Minocycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Glatiramer Acetate injection with oral minocycline (Active Comparator): Glatiramer Acetate 20mg with oral minocycline 100mg
  Interventions: Drug: glatiramer acetate with minocycline
- Glatiramer Acetate with placebo (Experimental): Glatiramer acetate injection 20mg with oral placebo
  Interventions: Drug: Glatiramer acetate with placebo

INTERVENTIONS:
Drug: glatiramer acetate with minocycline — Subcutaneous injection glatiramer acetate 20mg, with oral minocycline 100mg
  Other Names: Copaxone®
  Arms: Glatiramer Acetate injection with oral minocycline
Drug: Glatiramer acetate with placebo — Subcutaneous injection glatiramer acetate 20mg, with oral placebo
  Other Names: Copaxone®
  Arms: Glatiramer Acetate with placebo

SUMMARY:
This study investigates the add-on effect of oral minocycline in subjects treated with daily injection of Copaxone. Copaxone and minocycline are thought to have differential modes of actions that may complement each other in treating MS symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically definite MS as defined by Poser et al. (Ann. Neurol. 1983) with disease duration (from onset) of at least 6 months.
2. Subjects must have a relapsing-remitting disease course.
3. Subjects must have had at least 1 documented relapse within the last year prior to study entry.
4. Subjects must have at least 1 and not more than 15 gadolinium (Gd)-enhancing lesions on the screening MRI scan.
5. Subjects must be relapse-free and not have taken corticosteroids (IV, IM and/or PO) within the 30 days prior to the screening visit.
6. Subjects may be male or female. Women of child- bearing potential must use a contraceptive method deemed reliable by the investigator.
7. Subjects must be between the ages of 18 and 50 years inclusive.
8. Subjects must be ambulatory, with a Kurtzke EDSS score of between 0 and 5.0 inclusive.
9. Subjects must be willing and able to give written informed consent prior to entering the study.

Exclusion Criteria:

1. Previous use of injectable glatiramer acetate.
2. Previous use of cladribine.
3. Previous use of immunosuppressive agents in the last 6 months.
4. Use of experimental or investigational drugs, including I.V. immunoglobulin and statins, within 6 months prior to study entry.
5. Use of interferon agents or minocycline within 4 months prior to the screening visit.
6. Chronic corticosteroid (IV, IM and/or PO) treatment (more than 30 consecutive days) in the 6 months prior to study entry.
7. Previous total body irradiation or total lymphoid irradiation (TLI).
8. Pregnancy or breast feeding.
9. Subjects who experience a relapse between the screening (month -1) and baseline (month 0) visits.
10. Significant medical or psychiatric condition that affects the subject's ability to give informed consent, or to complete the study, or any condition which the investigator feels may interfere with participation in the study (e.g. alcohol or drug abuse).
11. A known history of sensitivity to mannitol.
12. Contraindication to or known history of sensitivity to tetracyclines.
13. A known history of sensitivity to gadolinium.
14. Inability to successfully undergo MRI scanning.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2004-06; Primary Completion 2006-06 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the add-on treatment effect of oral minocycline in subjects treated with daily injection of GA as reflected by number of MRI T1 Gd-enhancing lesions in T1-weighted images. | 24 months

SECONDARY OUTCOMES:
Assessment of tolerability and safety | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean Godin, MD, Study Director — Teva Neuroscience Canada

REFERENCES:
- [Result] Metz LM, Li D, Traboulsee A, Myles ML, Duquette P, Godin J, Constantin M, Yong VW; GA/minocycline study investigators. Glatiramer acetate in combination with minocycline in patients with relapsing--remitting multiple sclerosis: results of a Canadian, multicenter, double-blind, placebo-controlled trial. Mult Scler. 2009 Oct;15(10):1183-94. doi: 10.1177/1352458509106779. Epub 2009 Sep 23. PMID 19776092